CLINICAL TRIAL: NCT00887939
Title: Pathogenesis and Genetic Basis of Physical Induced Urticarial Syndromes
Brief Title: Pathogenesis of Physical Induced Urticarial Syndromes
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 090126; 09-I-0126
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-04-15

CONDITIONS: Hypersensitivity, Immediate; Autoinflammatory Syndromes; Physical Urticaria; Familial Cold Autoinflammatory Syndrome
Keywords: Hives; Inflammasome; Mast Cell; Natural History; Urticaria
MeSH Terms: conditions — Hypersensitivity, Immediate; Familial dermographism; Cryopyrin-Associated Periodic Syndromes; Urticaria

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Affected physical urticaria
- 2: Healthy volunteer
- 3: Unaffected relative

SUMMARY:
Background:

* Urticaria is a common itchy skin disorder that may occur spontaneously or on exposure to a physical trigger (called physical urticaria).
* Researchers are studying the genetic basis of a physically induced urticarial syndrome. Once called familial cold urticaria, this condition is now called familial cold autoinflammatory syndrome (FCAS). FCAS is an autoinflammatory disease, a group of inherited disorders characterized by unprovoked episodes of inflammation. Patients with FCAS often have hives, joint pain, and fever following general exposure to cold.
* Patients with FCAS have a mutation in a gene that makes a protein called cryopyrin. Cryopyrin seems to be involved with the production of a proinflammatory mediator called interleukin-1 (IL-1). Patients with FCAS and others with autoinflammatory syndromes have benefited from medication that blocks the effects of IL-1.

Objectives:

* To investigate mechanisms that may cause physical hives or urticaria.
* To reproduce urticaria through challenge testing (procedures to test the skin for a reaction to a stimulus), followed by mast cell studies, measurement of IL-1, genetic studies, and other molecular studies to lead to a better understanding of urticaria and to design safe and more effective treatments.

Eligibility:

* Patients between 6 months and 65 years of age with a documented history of clinically reproducible physical urticaria that triggers hives and that has been evaluated by a physician. Patients should have a letter of referral, including copies of pertinent medical history and laboratory studies, from a referring physician.
* Affected and nonaffected family members of such patients.
* Exclusion criteria include (1) the presence of conditions that may put the subject at undue risk, such as acute infection, severe thrombocytopenia (a lower than normal number of platelets in the blood), or significant cardiovascular disease; (2) any condition that would make the subject unsuitable for enrollment in this study; and (3) a history of HIV, other known immunodeficiency, or evidence of chronic Hepatitis B and/or C infection.

Design:

* Researchers will conduct the following tests to verify which triggers cause the hives:

  * History and physical exam to determine the relationship between the trigger and appearance of the hives.
  * Blood samples for baseline screening (additional samples may be taken within 8 hours of triggering hives).
  * Verification of hives using standard challenge testing.
* Procedures to trigger urticaria (the challenge testing) include dermatographism (stroking the skin), delayed pressure urticaria (direct pressure), cold-induced urticaria (cold exposure), cholinergic urticaria (exercise, hot water), solar urticaria (sun exposure), localized heat urticaria (direct heat exposure), aquagenic urticaria (room temperature water), and vibratory angioedema (direct vibratory stimulus exposure).
* Participants who have a positive history for hives and failed challenge testing (that is, hives resulted from the triggers) will be asked to provide a skin biopsy and additional bloods samples for research purposes.
* Participants will be asked to return to the clinic within 1 month if multiple triggers could not be verified during the initial visit, or to return for additional research evaluations, which may include a skin punch biopsy and blood sample collection. Patients may have to stay at the hospital overnight, if required to document the disease.
* Nonaffected family members who enroll in this protocol will provide samples for comparison with the family member who has a history of hives.
* Participants will receive a small financial compensation for the skin biopsy.

DETAILED DESCRIPTION:
Urticaria is a common skin disorder that is classified according to its chronicity into acute and chronic forms. It may occur spontaneously or on exposure to a physical factor. In the latter case, the urticaria is classified as a physical urticaria . Physical urticaria may be induced by mechanical and applied pressure, exercise, or exposure to cold, heat, sun, water, or vibration. The urticarial lesions are generally thought to be the result of mast cell activation and degranulation, which is supported by the finding of increased levels of serum histamine during some urticarial flares. Passive transfer experiments, whereupon serum from affected donors is transferred into recipient s skin followed by physical stimulation with resultant urticaria at the site of challenge, have been positive in some instances. This suggests the presence of an intrinsic factor in serum, such as IgE, which then mediates activation of tissue mast cells. However, the pathogenesis in general remains unclear and a genetic basis for these disorders has not been elucidated.

The goal of this protocol is thus to gain a better understanding of the pathogenesis of physical urticaria through the investigation of subjects with severe and unusual phenotypes and/or inherited patterns of disease. Subjects will undergo a clinical evaluation that will include verification of their urticaria. Blood and tissue samples, if available, will be collected for analysis. The analysis will be targeted toward the determination of novel serum mediators, mast cell activation and mutational analysis in families with inherited patterns.

ELIGIBILITY:
* INCLUSION CRITERIA:

Affected subjects/guardian must:

1. Be at least 2 years of age and no older than 90 years of age
2. Have a history of a physical urticaria, which has been evaluated by the patient's healthcare practitioner.
3. Provide copies of pertinent medical records and laboratory studies
4. Have a health care provider outside of NIH
5. Be willing to give informed consent
6. Be willing to donate blood for sample storage to be used for future research

Non-affected relatives/guardian must:

1. Be at least 2 years of age and no older than 90 years of age
2. Have a relative who is enrolled on this protocol and is known to have a documented history of a physical urticaria
3. Not have a history of physical urticaria
4. Be willing to give informed consent
5. Be willing to donate blood for sample storage to be used for future research

Healthy volunteers must:

1. Be 18-65 years of age
2. Be non-atopic (not have a history of allergic rhinitis, asthma, atopic dermatitis) per subject medical history
3. Have the ability to give informed consent
4. Be willing to donate blood for sample storage to be used for future research
5. Not have a history of physical urticaria

EXCLUSION CRITERIA:

The following criteria apply to all subjects:

1. Presence of conditions which, in the judgment of the investigator or the referring physician, may put the subject at undue risk, such as acute infection, severe thrombocytopenia (minimum platelet count of 30,000), or significant cardiovascular disease
2. Any condition that in the view of the principal investigator (PI) would make the subject unsuitable for enrollment in this study
3. History of HIV or other known immunodeficiency
4. History or evidence of chronic Hepatitis B and/or C infection
5. Pregnancy

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2009-06-17 (Actual)

PRIMARY OUTCOMES:
to determine the role of mast cell activation and genetic predisposition in the pathogenesis of physically induced urticaria. | 12/31/2028
  The patient s physical urticaria will be verified through standard testing.

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh D Komarow, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IDP will not be shared since sequencing is performed through NIH Centralized sequencing.

REFERENCES:
- [Background] Meyer J, Gorbach AM, Liu WM, Medic N, Young M, Nelson C, Arceo S, Desai A, Metcalfe DD, Komarow HD. Mast cell dependent vascular changes associated with an acute response to cold immersion in primary contact urticaria. PLoS One. 2013;8(2):e56773. doi: 10.1371/journal.pone.0056773. Epub 2013 Feb 22. PMID 23451084
- [Background] Boyden SE, Desai A, Cruse G, Young ML, Bolan HC, Scott LM, Eisch AR, Long RD, Lee CC, Satorius CL, Pakstis AJ, Olivera A, Mullikin JC, Chouery E, Megarbane A, Medlej-Hashim M, Kidd KK, Kastner DL, Metcalfe DD, Komarow HD. Vibratory Urticaria Associated with a Missense Variant in ADGRE2. N Engl J Med. 2016 Feb 18;374(7):656-63. doi: 10.1056/NEJMoa1500611. Epub 2016 Feb 3. PMID 26841242
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-I-0126.html